CLINICAL TRIAL: NCT05527041
Title: A Highly Portable Device for Assessment of Mild Traumatic Brain Injury in Deployed and Far-Forward Settings
Status: Enrolling by invitation | Type: Observational
Sponsor: Oculogica, Inc. (Industry)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: W81XWH21C0103
Record Dates: First submitted 2022-08-30; First posted 2022-09-02 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-03

CONDITIONS: Concussion, Brain; Mild Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Eye-tracking; Far-forward Settings; Return-to-Activity; Diagnostic
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Concussed: Subjects age 17-34 years within 72 hours of injury.
  Interventions: Device: EyeBOX Lens (EBLens)
- Non-concussed: In Phase I, uninjured, matched controls. In Phase II, subjects completing baseline concussion testing as part of the standard of care or athletics pre-season.
  Interventions: Device: EyeBOX Lens (EBLens)

INTERVENTIONS:
Device: EyeBOX Lens (EBLens) — The investigational device, EBLens, consists of eye-tracking scanners and sensors, developed by AdHawk Microsystems, embedded into a rugged pair of eye-glasses. The subject will wear the EBLens form factor while seated about 40 cm from a small handheld computer screen. The subject will be instructed to watch a video on the screen, while trying not to move their head. The operator will then initiate the EBLens test sequence. During this test a video will be displayed on only a portion of the screen (aperture about 1/9 the size of the screen) for 90 seconds. The video aperture will begin in the upper left corner, and, after 10 seconds, moves in a clockwise direction around the screen for 2 cycles, each taking 40 seconds. During the scan, the following data are collected at a frame rate from 100 to 500 Hz:
  * Gaze coordinates
  * Pupil sizes
  * Accelerometer data
  * Gyroscopic data
  * Rotation data
  * Blink data

SUMMARY:
The purpose of this study is to develop a highly portable, ruggedized diagnostic tool for concussion, EyeBOX Lens (EBLens), that can be utilized in deployed field and far-forward settings. The EBLens will be based on a concussion diagnostic algorithm from the FDA cleared EyeBOX device, developed by Oculogica, and eye-tracking data collected from a wearable set of eye-tracking glasses, developed by Adhawk Microsystems. Once the EBLens is prototyped, an algorithm for diagnosing concussion will be developed that is specifically appropriate for the EBLens via a case-control clinical study comparing 100 concussed to 100 non-concussed subjects (Phase I). Participants, age 18-35 years, will be recruited from the KACH research team and affiliated providers and clinical sites. Concussed individuals will be assessed within 72 hours of concussion. Demographics, basic medical history, symptom severity, a visio-vestibular exam and the EBLens scan will be collected on both injured cases and uninjured controls at a single time point.

The algorithm and the EBLens will be validated in a subsequent, prospective cohort validation study (Phase II) designed for FDA submission. The correlation of the EBLens output with resolution of symptoms will also be observed in longitudinal follow-up of concussed participants in the validation study. The participant population for this study will be cadets recruited from the USMA and young athletes recruited from affiliated sites during baseline concussion testing. Participants will be assessed at baseline at the start of their academic year or sports season. Those participants who experience a concussive injury will be assessed again at three time points; 1) within 72 hours of injury, 2) weekly until and at the time of initiation of a graded return to activity protocol, and 3) upon clearance for unrestricted RTP/RTD.

ELIGIBILITY:
CONCUSSED:

Inclusion Criteria:

* Provide documented informed consent.
* Have presented, at any time post injury, for any complaint related to an injury involving either a direct force to the head or a blow to the body that has the potential to transmit a rapid acceleration/deceleration of the head, with or without loss of consciousness, with or without external signs of head injury.
* Be a current cadet/enrolled student age 17-34.
* Have the ability to provide a complete ophthalmologic, medical, and neurologic history as well as report current medications.

Exclusion Criteria:

* Have penetrating trauma or known skull fracture or intracranial injury.
* Have had a conventional head CT or MRI demonstrating evidence of structural brain injury (subdural, epidural or intraparenchymal hemorrhage, edema/mass effect per attending radiologist read).
* Be blind (no light perception), have missing or non-functional eyes.
* Be unable to open their eyes.
* Have a history of unresolved strabismus, diplopia, amblyopia.
* Have a history of unresolved cranial nerve III, IV, or VI palsy.
* Have a history of unresolved macular edema, retinal degeneration, extensive cataract, or ocular globe disruption.
* Have a history of extensive prior eye surgery or scarring (examples include strabismus surgery, scleral buckle repair of retinal detachment, repair of blow out fractures of the orbit and any procedures that would interfere with extraocular muscle movements; prior cataract surgery or Lasik are not exclusions).
* Have a prior history of unresolved ocular-motor dysfunctions.
* Be intoxicated.

CONTROLS:

Inclusion Criteria:

* Provide documented informed consent.
* Be a current cadet/enrolled student age 17-34.
* Have the ability to provide a complete ophthalmologic, medical, and neurologic history as well as report current medications.

Exclusion Criteria:

* Have presented, within the prior six months, for any complaint related to an injury involving either a direct force to the head or a blow to the body that has the potential to transmit a rapid acceleration/deceleration of the head, with or without loss of consciousness, with or without external signs of head injury.
* Have penetrating trauma or known skull fracture or intracranial injury.
* Have had a conventional head CT or MRI demonstrating evidence of structural brain injury (subdural, epidural or intraparenchymal hemorrhage, edema/mass effect per attending radiologist read).
* Be blind (no light perception), have missing or non-functional eyes.
* Be unable to open their eyes.
* Have a history of unresolved strabismus, diplopia, amblyopia.
* Have a history of unresolved cranial nerve III, IV, or VI palsy.
* Have a history of unresolved macular edema, retinal degeneration, extensive cataract, or ocular globe disruption.
* Have a history of extensive prior eye surgery or scarring (examples include strabismus surgery, scleral buckle repair of retinal detachment, repair of blow out fractures of the orbit and any procedures that would interfere with extraocular muscle movements; prior cataract surgery or Lasik are not exclusions).
* Have a prior history of unresolved ocular-motor dysfunctions.
* Be intoxicated.

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants will be young athletes or cadets between the ages of 18-35. Cadets at the USMA who are 17 and are emancipated will also be included. To be included in the algorithm development study, subjects must either be uninjured (to fall into the uninjured cohort) or have experienced a concussive event (to fall into the injured cohort). In the validation study, subjects must be participants who have completed baseline testing and have consented to participate.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-26 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of acute clinical diagnosis of concussion using EBLens form factor and algorithm | Within 72 hours of injury
  The EBLens will have at least 70% sensitivity and specificity for diagnosis of acute concussion

SECONDARY OUTCOMES:
Diagnostic accuracy of recovery determination for return to activity and duty (RTA / RTD) using EBLens form factor and algorithm | Through study completion, up to one year
  The EBLens will have at least 70% sensitivity and specificity for recovery determination for return to activity and duty (RTA / RTD) without complication.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Cameron, PhD, Principal Investigator — Keller Army Community Hospital; Christina Master, MD, Principal Investigator — Children's Hospital of Philadelphia; Sadie Buboltz-Dubs, PhD, Principal Investigator — University of Wisconsin - Green Bay
Locations (1):
- Keller Army Hospital, West Point, New York, United States